CLINICAL TRIAL: NCT00063687
Title: A Phase II-III Prospective, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Oxypurinol Added to Standard Therapy in Patients With NYHA Class III-IV Congestive Heart Failure
Brief Title: Oxypurinol Compared With Placebo for Class III-IV NYHA Congestive Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 500-02-01
Record Dates: First submitted 2003-07-02; First posted 2003-07-03 (Estimated); Last update posted 2005-08-05 (Estimated); Status verified 2003-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Oxypurinol

INTERVENTIONS:
Drug: Oxypurinol

SUMMARY:
The OPT-CHF (OxyPurinol Therapy for CHF) study is designed to demonstrate the efficacy and safety of oral oxypurinol vs. placebo in a randomized, double-blind, twenty-four week trial in 400 patients in up to 50 centers. Measures of clinical efficacy (NYHA class and Patient Global Assessment) as well as clinical outcomes (e.g., death, worsening heart failure, and hospitalization) will be assessed as a composite endpoint in this trial.

ELIGIBILITY:
Inclusion criteria

* 18-85 years old,
* Stable NYHA Class III-IV
* Hospitalization or ER visits in past 18 months for worsening Heart Failure (or addition of new heart failure medication added to regimen due to lack of stability on current regimen.
* EF =< 40%

Exclusion criteria

* Any condition (other than CHF) that could limit exercise
* Any concurrent disease likely to limit life expectancy.
* Participation in another clinical trial
* Primary valvular disease, active myocarditis, or an obstructive or restrictive cardio-myopathy
* Heart Attack, Stroke, Unstable Angina or Cardiac surgery within previous 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-03; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hare, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Carr-Dzindzio Cardiology, Oceanside, California
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Saint Vincents Hospital and Medical Center, New York, New York

REFERENCES:
- [Derived] Hare JM, Mangal B, Brown J, Fisher C Jr, Freudenberger R, Colucci WS, Mann DL, Liu P, Givertz MM, Schwarz RP; OPT-CHF Investigators. Impact of oxypurinol in patients with symptomatic heart failure. Results of the OPT-CHF study. J Am Coll Cardiol. 2008 Jun 17;51(24):2301-9. doi: 10.1016/j.jacc.2008.01.068. PMID 18549913
- See also: Related Info — http://www.cardiome.com